CLINICAL TRIAL: NCT02184572
Title: Safety and Immunogenicity Study of GSK Biologicals' Measles-mumps-rubella (MMR) Vaccine (209762) Comparing Immunogenicity and Safety to Merck & Co., Inc.'s MMR Vaccine, in Healthy Children 12 to 15 Months of Age
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' Measles, Mumps and Rubella (MMR) Vaccine (209762) Compared to Merck & Co., Inc.'s MMR Vaccine in Healthy Children 12 to 15 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115650; 2011-006161-18 (EudraCT Number)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Measles; Mumps; Rubella; Measles-Mumps-Rubella Vaccine
Keywords: Rubella; Healthy children; Measles; Safety; Mumps; 12 to 15 months; Immunogenicity
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine; Vaccines; Chickenpox Vaccine; Hepatitis A Vaccines; 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- INV_MMR (Experimental): Subjects receive 1 dose of the study vaccine Priorix co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also receive Prevnar 13 at Day 0.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- COM_MMR (Active Comparator): Subjects receive 1 dose of the licensed vaccine M-M-R II or M-M-R VaxPro Lot 1 or Lot 2 co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also receive Prevnar 13 at Day 0.
  Interventions: Biological: M-M-R II; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13

INTERVENTIONS:
Biological: Priorix — 1 dose administered subcutaneously in the triceps region of left arm at Day 0
  Other Names: GSK Biologicals' live attenuated measles; mumps and rubella (MMR) vaccine
  Arms: INV_MMR
Biological: M-M-R II — 1 dose administered subcutaneously in the triceps region of left arm at Day 0
  Other Names: MMR vaccine live (M-M R II; Merck & Co.; Inc.; or M-M-R VaxPro; Sanofi Pasteur/Merck Sharp and Dohme [SPMSD])
  Arms: COM_MMR
Biological: Varivax — 1 dose administered subcutaneously in the triceps region of right arm at Day 0
  Other Names: Merck & Co. Inc.'s Varicella virus vaccine; live
Biological: Havrix — 1 dose administered intramuscularly in the anterolateral region of the right thigh at Day 0
  Other Names: GSK Biologicals' Hepatitis A vaccine; inactivated
Biological: Prevnar 13 — 1 dose administered intramuscularly in the anterolateral region of the left thigh at Day 0 to subjects recruited in US
  Other Names: Pfizer Inc.'s Pneumococcal 13-valent conjugate vaccine (diphtheria CRM197 protein)

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' trivalent MMR (Priorix), comparing it to Merck's MMR vaccine (M-M-R II), which is approved for use in the US in healthy children 12 to 15 months of age.

DETAILED DESCRIPTION:
This study will evaluate the safety of GSK's trivalent MMR vaccine (referred to as INV_MMR vaccine) at a potency that will be used to define maximum release limits for the INV_MMR in comparison to the US standard of care (M-M-R II/ M-M-R VaxPro vaccine referred to as COM_MMR vaccine). In order to obtain more representative data on the comparator vaccine, the COM_MMR used in this study will consist of two lots designated COM_MMR_L1 and COM_MMR_L2. Throughout the study COM_MMR_L1 and COM_MMR_L2 will be analyzed as pooled lots. This study is intended to support licensure of GSK's MMR vaccine in the US.

All children will receive Varivax and Havrix vaccines, concomitantly with MMR containing vaccine at 12 to 15 months of age. Prevnar 13 will be administered only to US children. At the end of the study, GSK will provide a second dose of Havrix and/or varicella vaccine to participants enrolled in selected non-US countries if local health departments do not routinely provide hepatitis A and varicella vaccination. The second dose of Havrix and varicella vaccine is not part of the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child between 12 and 15 months of age (e.g., from the 1 year birthday until the day before age 16 months) at the time of vaccination.
* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the child.
* Child is in stable health as determined by investigator's clinical examination and assessment of child's medical history.
* For US children only: a child who received all routine vaccinations as per ACIP recommendations prior to study entry: completion of hepatitis B and rotavirus series and completion of the primary series of diphtheria, tetanus, pertussis, poliovirus, Haemophilus influenzae type b (Hib) and pneumococcal vaccines. The 3-dose infant series of Prevnar 13 should be completed at least 60 days prior to study vaccination.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) during the period starting 30 days before the day of study vaccination (i.e., 30 days prior to Day 0) or planned use during the entire study period.
* Concurrently participating in another clinical study, in which the child has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration (defined as 14 or more consecutive days) of immunosuppressants, or other immune-modifying drugs during the period starting 180 days prior to the study vaccination at Visit 1 or any planned administration of immunosuppressive and immune-modifying drugs during the entire study.

  * For corticosteroids, this will mean prednisone ≥0.5 mg/kg/day or equivalent.
  * Inhaled and topical steroids are allowed.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days prior to the day of study vaccination at Visit 1 and ending at Visit 2. Please Note:

  * Inactivated influenza (Flu) vaccine and monovalent Haemophilus influenzae type b conjugate vaccine (Hib) vaccines may be given at any time, including the day of study vaccination (Flu and Hib vaccines must be administered at a different location than the study vaccine/s).
  * Any other age appropriate vaccine may be given starting at Visit 2 and anytime thereafter.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days before the study vaccination at Visit 1 or planned administration from the date of vaccination through the immunogenicity evaluation at Visit 2.
* History of measles, mumps, rubella, varicella/zoster and/or hepatitis A disease.
* Known exposure to measles, mumps, rubella and/or varicella/zoster during the period starting within 30 days prior to first study vaccination.
* Previous vaccination against measles, mumps, rubella, hepatitis A and/or varicella virus.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including hypersensitivity to neomycin, latex or gelatin.
* Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever). Fever is defined as temperature ≥38.0°C/100.4°F by any age appropriate route. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection without fever.
* Active untreated tuberculosis based on medical history.
* Any other condition which, in the opinion of the investigator, prevents the child from participating in the study.
* For US children only: a child that previously received a fourth dose of PCV-13 vaccine.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1742 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (72):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Baldwin Park, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Mandan, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Cheraw, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Watertown, South Dakota
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, League City, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Payson, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Ellensburg, Washington
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
  - GSK Investigational Site, Monroe, Wisconsin
- GSK Investigational Site, Tartu, Estonia
- Finland (5):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Puerto Rico (3):
  - GSK Investigational Site, Guayama
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

REFERENCES:
- [Background] MMR-162 Study Group. Safety and immunogenicity of an upper-range release titer measles-mumps-rubella vaccine in children vaccinated at 12 to 15 months of age: a phase III, randomized study. Hum Vaccin Immunother. 2018;14(12):2921-2931. doi: 10.1080/21645515.2018.1502527. Epub 2018 Aug 29. PMID 30118386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 subjects from 1742 were allocated subject number but no study vaccine was administered. Therefore, the number of subjects started in 1736.
Pre-assignment Details: US sub-cohort: Subjects recruited in US received INV_MMR (Priorix) or COM_MMR (M-M-R II/M-M-R VaxPro) co-administered with Varivax, Havrix & Prevnar 13 vaccines (Day 0). Non-US sub-cohort: Subjects recruited outside the US received INV_MMR (Priorix) or COM_MMR (M-M-R II/M-M-R VaxPro) co-administered with Varivax & Havrix vaccines (Day 0).
Groups:
- INV_MMR: Subjects received 1 dose of the study vaccine Priorix co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also received Prevnar 13 at Day 0.
- COM_MMR: Subjects received 1 dose of the licensed vaccine M-M-R II or M-M-R VaxPro Lot 1 or Lot 2 co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also received Prevnar 13 at Day 0.
Period: Overall Study
Arm/Group | INV_MMR | COM_MMR
Started | 1164 | 572
Completed | 1117 | 542
Not Completed | 47 | 30
Not completed — Lost to Follow-up | 29 | 21
Not completed — Family Out Of Country Until 9/29/2015 | 1 | 0
Not completed — Loss Of Kaiser Insurance | 1 | 0
Not completed — 2nd blooddraw & diary card incomplete | 1 | 0
Not completed — Traveling Outside The Country | 1 | 0
Not completed — Withdrawal by Subject | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INV_MMR | COM_MMR | Total
Number analyzed (Participants) | 1164 | 572 | 1736
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.3 (0.7) | 12.3 (0.7) | 12.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 551 | 270 | 821
  Male | 613 | 302 | 915
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage / African American | 64 | 38 | 102
  American Indian or Alaskan Native | 29 | 16 | 45
  Asian - Central/South Asian Heritage | 9 | 4 | 13
  Asian - East Asian Heritage | 131 | 65 | 196
  Asian - Japanese Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 28 | 12 | 40
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White - Arabic / North African Heritage | 3 | 3 | 6
  White - Caucasian / European Heritage | 808 | 385 | 1193
  Other | 89 | 47 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever After MMR (Priorix or M-M-R II/M-M-R VaxPro [Lot 1 or Lot 2]) Vaccination
Description: Fever was assessed for temperature equal to/above (≥) 38.0°C and above (>) 39.0°C. The safety profile for fever was assessed based on the group difference (INV_MMR minus COM_MMR) in incidence of fever equal to or below the cut-off value.
Time Frame: During Day 5 to Day 12 post-vaccination period
Population: Analysis was performed on Total Vaccinated cohort (TVC) which included all vaccinated subjects with administration of either Priorix or M-M-R II/M-M-R VaxPro lots documented.
Measure: Count of Participants; unit: Participants
Groups:
- INV_MMR Group: Subjects received 1 dose of the study vaccine Priorix co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also received Prevnar 13 at Day 0.
- COM_MMR Group: Subjects received 1 dose of the licensed vaccine M-M-R II or M-M-R VaxPro Lot 1 or Lot 2 co-administered with Varivax and Havrix vaccines at Day 0. Subjects recruited in the US also received Prevnar 13 at Day 0.
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1126 | 555
Participants
  > 39.0°C | 47 | 17
  ≥ 38.0°C | 205 | 95
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Difference between groups (INV_MMR Group minus COM_MMR Group) in incidence of fever > 39.0°C; Test type: Non-Inferiority or Equivalence — The upper limit of the 2-sided standardised asymptotic 95% Confidence Interval (CI) for the group difference (INV_MMR minus COM_MMR) in incidence of fever ≥ 39.0°C (≥ 102.2°F) should be equal to or below 5%; Difference in incidence of fever = 1.11, 95% CI 2-sided [-0.93 to 2.89]
Statistical Analysis 2: Comparison: INV_MMR Group vs COM_MMR Group; Difference between groups (INV_MMR Group minus COM_MMR Group) in incidence of fever > 38.0°C; Test type: Non-Inferiority or Equivalence — The upper limit of the 2-sided standardised asymptotic 95% CI for the group difference (INV_MMR minus COM_MMR) in incidence of fever ≥ 38.0°C (≥ 100.4°F) should be equal to or below 10%; Difference in incidence of fever = 1.09, 95% CI 2-sided [-2.89 to 4.85]

2. Secondary Outcome: Percentage of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-measles virus antibody concentration greater than or equal to [≥] 200 milli International Units per milliliter [mIU/mL] (Enzyme-Linked Immunosorbent Assay [ELISA], Enzygnost) among subjects who were seronegative (antibody concentration less than [<] 150 mIU/mL) before vaccination.
Time Frame: At Day 42 post vaccination
Population: According to Protocol (ATP) cohort for immunogenicity: included all eligible subjects with pre and post-vaccination serology results available for at least one vaccine components of measles, mumps or rubella, who did not meet any elimination criteria up to the Visit 2 blood sample and who complied with the post dose blood sample schedule.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1043 | 521
Percentage of subjects
  ≥ 150 mIU/mL | 99.3 [98.6 to 99.7] | 96.7 [94.8 to 98.1]
  ≥ 200 mIU/mL | 99.0 [98.2 to 99.5] | 96.5 [94.6 to 97.9]

3. Secondary Outcome: Anti-measles Virus Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. Analyses included initially seronegative subjects only.
Time Frame: At Day 42 post vaccination
Population: ATP cohort for immunogenicity: included all eligible subjects with pre and post-vaccination serology results available for at least one vaccine components of measles, mumps or rubella, who did not meet any elimination criteria up to the Visit 2 blood sample and who complied with the post dose blood sample schedule.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1043 | 521
mIU/mL | 2751.9 [2618.3 to 2892.2] | 3133.3 [2878.6 to 3410.6]

4. Secondary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥ 10 ELISA Unit per milliliter [EU/mL] (ELISA, Pharmaceutical Product Development, Inc.[PPD]) among subjects who were seronegative (antibody concentration < 5 EU/mL) before vaccination.
Time Frame: At Day 42 post vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 964 | 483
Percentage of subjects
  ≥ 5 EU/mL | 99.8 [99.3 to 100] | 99.4 [98.2 to 99.9]
  ≥ 10 EU/mL | 99.4 [98.7 to 99.8] | 97.9 [96.2 to 99.0]

5. Secondary Outcome: Anti-mumps Virus Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in EU/mL. Analyses included initially seronegative subjects only.
Time Frame: At Day 42 post vaccination
Population: According to Protocol (ATP) cohort for immunogenicity: included all eligible subjects with pre and post-vaccination serology results available for at least one vaccine components of measles, mumps, or rubella, who did not meet any elimination criteria up to the Visit 2 blood sample and who complied with the post dose blood sample schedule.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 964 | 483
EU/mL | 86.0 [82.0 to 90.3] | 82.6 [76.5 to 89.2]

6. Secondary Outcome: Percentage of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥ 10 International Unit per milliliter [IU/mL] (ELISA, Enzygnost) among subjects who were seronegative (antibody concentration < 4 IU/mL) before vaccination.
Time Frame: At Day 42 post vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1043 | 521
Percentage of subjects
  ≥4 IU/mL | 99.6 [99.0 to 99.9] | 99.8 [98.9 to 100]
  ≥10 IU/mL | 95.7 [94.3 to 96.8] | 98.3 [96.7 to 99.2]

7. Secondary Outcome: Anti-rubella Virus Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in IU/mL. Analyses included initially seronegative subjects only.
Time Frame: At Day 42 post vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1043 | 521
IU/mL | 45.0 [42.8 to 47.2] | 66.8 [62.3 to 71.7]

8. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed solicited local AEs were injection site pain, redness and swelling. Any = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on TVC which included all vaccinated subjects with administration of either Priorix or M-M-R II/M-M-R VaxPro lots documented.
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1123 | 553
Participants
  Any pain | 312 | 131
  Any redness (mm) | 260 | 137
  Any swelling (mm) | 96 | 58

9. Secondary Outcome: Number of Subjects With Any Solicited General AEs
Description: Assessed solicited general AEs were drowsiness, irritability/fussiness and loss of appetite. Any = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 15-day (Days 0-14) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1126 | 555
Participants
  Any drowsiness | 527 | 238
  Any irritability/fussiness | 722 | 345
  Any loss of appetite | 493 | 232

10. Secondary Outcome: Number of Subjects Reporting Any Fever
Description: Any fever (≥ 38°C) = Occurrence of fever regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1126 | 555
Participants | 350 | 179

11. Secondary Outcome: Number of Subjects Reporting Any Rash
Description: Any rash = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1126 | 555
Participants
  Any localized or generalized | 275 | 152
  Any with fever | 100 | 48
  Any varicella like | 40 | 22
  Any measles/rubella like | 65 | 26

12. Secondary Outcome: Number of Subjects Reporting MMR Specific Solicited General AEs
Description: Assessed MMR specific solicited general AEs were parotid gland swelling and any suspected signs of meningism including febrile convulsions. Any = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1126 | 555
Participants
  Any parotid gland swelling | 0 | 0
  Any febrile convulsion | 2 | 0

13. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Unsolicited AE included any AE reported in addition to those solicited during the clinical study and any 'solicited' AE with onset outside the specified period of follow-up for solicited AEs. Any = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1164 | 572
Participants | 598 | 277

14. Secondary Outcome: Number of Subjects Reporting AEs of Specific Interest
Description: AEs of specific interest included new onset chronic disease (NOCD) (e.g., autoimmune disorders, asthma, type I diabetes, vasculitis, celiac disease, conditions associated with sub-acute or chronic thrombocytopenia and allergies) and AEs prompting emergency room (ER) visits.
Time Frame: Day 0 through the end of the study (Day 180)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1164 | 572
Participants
  NOCDs | 29 | 11
  AEs prompting ER visits | 166 | 55

15. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAE included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity. Any = Occurrence of AE regardless of intensity grade or relation to vaccination.
Time Frame: Day 0 through the end of the study (Day 180)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR | COM_MMR
Number analyzed (Participants) | 1164 | 572
Participants | 24 | 9

16. Secondary Outcome: Number of Subjects Reporting Measles-like Illness
Description: Measles-like illness was defined as the occurrence of the following signs/symptoms in the absence of another confirmed diagnosis:
  maculopapular rash (includes measles/rubella-like rash), fever (≥ 38°C) and at least one of the symptoms: cough, coryza (runny nose), conjunctivitis or diarrhea, with fever or rash. Other event must be one of cough, coryza, conjunctivitis, or diarrhea.
Time Frame: During Day 5 to Day 12 post-vaccination period
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 1164 | 572
Participants
  Measles-like illness | 18 | 5
  Maculopapular rash plus fever and one other event | 26 | 9
  Maculopapular rash and fever | 90 | 43

ADVERSE EVENTS:
Time Frame: SAEs = From Day 0 to study end (Day 180); Solicited local and general AEs = During the 4-day (Day 0-3) and 15-day (Day 0-14) post vaccination period, respectively; Unsolicited adverse events = During the 43-day (Day 0-42) post vaccination period.
Arm/Group | INV_MMR Group | COM_MMR Group
All-Cause Mortality (participants affected / at risk) | 0/1164 | 0/572
Serious Adverse Events (participants affected / at risk) | 24/1164 | 9/572
Other Adverse Events (participants affected / at risk) | 980/1164 | 477/572
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR Group (N=1164) | COM_MMR Group (N=572)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR Group (N=1164) | COM_MMR Group (N=572)
Diarrhoea (Gastrointestinal disorders) | 95 (105) | 46 (53)
Teething (Gastrointestinal disorders) | 59 (71) | 15 (17)
Injection site erythema (General disorders) | 284 (297) | 143 (149)
Injection site pain (General disorders) | 313 (314) | 133 (133)
Injection site swelling (General disorders) | 105 (108) | 61 (62)
Pyrexia (General disorders) | 350 (350) | 180 (180)
Otitis media (Infections and infestations) | 86 (95) | 35 (36)
Upper respiratory tract infection (Infections and infestations) | 111 (119) | 73 (75)
Decreased appetite (Metabolism and nutrition disorders) | 495 (497) | 233 (234)
Somnolence (Nervous system disorders) | 529 (529) | 238 (238)
Irritability (Psychiatric disorders) | 723 (740) | 348 (350)
Cough (Respiratory, thoracic and mediastinal disorders) | 80 (85) | 30 (31)
Rash (Skin and subcutaneous tissue disorders) | 275 (275) | 152 (152)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.